CLINICAL TRIAL: NCT04213144
Title: Randomized Double Blind Controlled Prospective Study to Evaluate the Influence of Electromagnetic Field as an Adjunctive Non Surgical Treatment in Implant With Peri-implantitis
Brief Title: Evaluate the Influence of Electromagnetic Field as an Adjunctive Non Surgical Treatment in Implant With Peri-implantitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, Hadar Zigdon MD, Rambam Health Care Campus, Rambam Health Care Campus
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0402-19-RMB CTIL
Record Dates: First submitted 2019-12-25; First posted 2019-12-30 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-04

CONDITIONS: Peri-Implantitis
MeSH Terms: conditions — Peri-Implantitis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Magdent Cap MED (Experimental): Soft and hard tissue healing with electomagnetic healing abutment.
  Interventions: Device: Magdent Cap MED
- Sham MED (Sham Comparator): Soft and hard tissue healing with a regular healing abutment.
  Interventions: Device: Sham MED

INTERVENTIONS:
Device: Magdent Cap MED — Magdent is intended to be used for accelaration of soft tissue and bone healing
  Arms: Magdent Cap MED
Device: Sham MED — Sham MED is intended to be used for soft tissue healing
  Arms: Sham MED

SUMMARY:
the aim of the study is to compare between two non-surgical methods of treatment of peri-implantitis by using debridement and placing an healing abutment with electomagnetic field (MED-Magdent Miniaturized Device) in the test group and Sham healing abutment in the control group ( Sham MED).

DETAILED DESCRIPTION:
Dental Implants are common alternative for replacement at the time of tooth loss. The two common methods for treatment implant with inflammation include surgical and global non-surgical treatment.

The non-surgical treatment includes soft tissue debridement with various tools which including manual, ultrasonic rotators, lasers and delayed release devices.

Using an electromagnetic field to induce bony healing in fractures and around implants is being investigated for studies and was found to be effective and safe. The electric field lowers osteoclasts activity, speeds up osteoid construction and stimulates creation blood vessels development. Forty patients who will attend to the department of periodontology at Rambam health care campus, at the School ofpostgraduate Dentistry, which will meet the research criteria, will be recruited. All patients will exhibit a moderate-onset gum infection around one of the implants.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent.
* Patients of 20 - 85 years.
* pocket depth of 5-8 mm and bone loss of 3-5mm Patients with fixed prosthodontics Implant with standart width

Exclusion Criteria:

* Heavy smokers (more than 10 cigarettes per day).
* Pregnant women
* active periodontal disease
* Consumption of Non Steroidal Anti Inflammatory drugs

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2020-03-03 (Actual); Primary Completion 2022-10-19 (Actual); Study Completion 2022-10-19 (Actual)

PRIMARY OUTCOMES:
Change in the implant probing depth (IPD) | baseline, 4 weeks, 12 weeks
  clinical measurement of the depth of the pocket around the implant in 6 sites

SECONDARY OUTCOMES:
changing in the concentration of the RANKL cytokine | baseline, 2 weeks, 4 weeks, 12 weeks
  Sampling the amount bycollecting gingival fluid with paper pins and examining the amount of the cytokine with ELISA (Enzyme Linked Immunoflorecance assay)asay

CONTACTS AND LOCATIONS:
Overall Officials: Hadar Zigdon, DMD, Principal Investigator — Rambam Health Care Campus
Locations (1):
- Rambam Health Care Campus, Dept. of Periodontology, Haifa, Israel